CLINICAL TRIAL: NCT01115114
Title: Treatment of Metabolic Syndrome in a Community Mental Health Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSC20090135H; 5R24MH072830 (NIH)
Record Dates: First submitted 2010-04-28; First posted 2010-05-04 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Serious Mental Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment as Usual (TAU) (Placebo Comparator): Study Intervention 1 Treatment as usual (TAU) will be psychiatry follow-up at local Community Mental Health Clinic at least every 3 months.
  Interventions: Behavioral: TAU
- IMBED (Active Comparator): Study Intervention 2 A Primary Care Provider (PCP) will be located within the community mental health clinic one day weekly to specifically run a Metabolic Syndrome Clinic.
  Interventions: Behavioral: IMBED
- Liaison (Active Comparator): Study Intervention 3 A Medical Case Manager(MCM) will be assigned to a patient who is identified on the basis of routine screening to need medical follow-up for metabolic syndrome.
  Interventions: Behavioral: Liaison

INTERVENTIONS:
Behavioral: TAU — A medical assistant will provide feedback on and educational materials describing the meaning of lab values to individuals identified as needing follow-up for metabolic syndrome, and will provide educational materials regarding healthy eating and exercise. The psychiatrist will recommend that the individual contact a primary care physician to follow-up on out of range values, and alter behaviors (over eating, being sedentary) to help improve health.
  Arms: Treatment as Usual (TAU)
Behavioral: IMBED — After identifying individuals through routine screening that need medical follow-up for metabolic syndrome, these individuals will be scheduled to see the on site primary care provider. Rapid scheduling (within 2 weeks) will be attempted. Patients will be seen by the primary care provider monthly or as needed as determined per patient. The primary care provider will prescribe medications for metabolic syndrome, discuss the patient with psychiatry staff and recommend follow-up appointments for physical problems based upon recommended guidelines and clinical judgment of necessity and urgency. Referral to a specialist will be made according to standard primary care practice guidelines. During the Metabolic Syndrome Clinic, if individuals bring up other medical conditions, they will be referred for treatment of these conditions to an outside primary care provider.
  Arms: IMBED
Behavioral: Liaison — Patients will be seen by the MCM bi-weekly or as needed as determined per patient. The MCM will discuss findings of the labs with the patient, work to get the individual an appointment with a primary care doctor, get releases of information to discuss treatment coordination between the primary care and psychiatric teams, obtain necessary records from primary care, and communicate findings to the treating psychiatrist. The MCM will also assist the patient in getting to primary care appointments by providing bus passes or other transportation, and with obtaining medications prescribed by the primary care provider. This may necessitate enrolling the patient in specific care plans as needed.
  Arms: Liaison

SUMMARY:
The purpose of this study is to learn if patients being treated with second generation antipsychotics and with clinically meaningful elevations/levels in any metabolic syndrome elements will have better access to medical treatment more quickly if they are randomized to one of the following conditions: 1) a primary care provider located in the community mental health center where mental health treatment is provided (IMBED), 2) a medical care manager to help coordinate treatment with an outside primary care provider (Liaison) or 3) the standard practice of advising the patient to see a primary care doctor (Treatment as Usual).

DETAILED DESCRIPTION:
Individuals will be identified for participation based upon baseline laboratory values obtained at the local Community Mental Health Clinic (CMHC) as part of the standard monitoring procedures for individuals on Second Generation Antipsychotics (SGAs). Following randomization, a research assistant will be assigned to obtain information on primary care provider visits, medications and lab tests conducted outside of the CMHC using a signed release for from the patient. Variables collected include: date and time of all physician or practitioner visits, type of practitioner, all medication prescriptions, and all laboratory values and vital signs related to metabolic syndrome parameters. Data will be put into an access data base for analysis. Data from private pharmacies will be obtained using a separate signed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18 years and older
* Active CMHC consumers
* Currently taking an atypical antipsychotic
* Identified as having clinically meaningful elevations/levels in metabolic indicators; i.e. fasting blood glucose (≥ 110), HDL ≤ 40mg/dl for males or ≤ 50mg/dl for females, blood pressure (≥ 130/85)
* Able to give informed consent
* Recipient of private or publicly-financed health insurance that includes medication coverage

Exclusion Criteria:

* Legally declared mentally incompetent (guardians will not be approached about study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Utilization of Care | 9 months
  We will compare the efficacy of IMBED, Liaison and Treatment as Usual for improving utilization of care. The primary outcome variables are time to contact with primary care practitioner, number of primary care visits, receiving appropriate medications, receiving appropriate labs, and receiving dietary and life style counseling.

SECONDARY OUTCOMES:
Metabolic Indicators | 9 months
  We will compare the efficacy of IMBED, Liaison and Treatment as Usual for improving metabolic indicators. The targets are biological variables measured over time (triglycerides, glucose, blood pressure, HDL, BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn I Velligan, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Center for Health Care Services, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas